CLINICAL TRIAL: NCT06578806
Title: Tooth Loss Rate and Its Associated Factors in Adult Population: a Retrospective Cross-sectional Study With up to 50 Years of Follow-up.
Brief Title: Tooth Loss Rate and Its Associated Factors: a Retrospective Cross-sectional Study With up to 50 Years of Follow-up.
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: USJ-2023-61
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Tooth Loss
Keywords: active therapy; bruxism; cardiovascular disease; diabetes; periodontitis; smoking; supportive periodontal therapy; tooth loss; tooth loss rate
MeSH Terms: conditions — Tooth Loss; Bruxism; Cardiovascular Diseases; Diabetes Mellitus; Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate, in an adult population (n=448) previously diagnosed with gingivitis and/ or periodontitis, the tooth loss rate and its potential associated factors such as diabetes, smoking, bruxism, cardiovascular diseases, and also the effect of supportive periodontal therapy on these factors, with an up to 50 years of follow-up period.

Significant results of the present study will help in the future reduction of tooth loss among periodontally involved patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years.
* Patients diagnosed with generalized chronic periodontitis or gingivitis.
* At least 10 years of follow-up after 1st visit.
* All treatments and recall sessions were done by the same operator at the same specialized dental clinic.

Exclusion Criteria:

* Patients with healthy periodontal status.
* Patients with orofacial anomalies and syndromes.
* Patients receiving periodontal treatments by different operators.
* Patients receiving periodontal treatments at different clinics.
* Patients receiving bisphosphonate therapy.
* Patients receiving chemotherapy or radiotherapy.
* Patients receiving a hormonal therapy.
* Patients with a history of refractory periodontitis or repeated abscess formation.
* Patients with debilitating diseases that could impair the immune system (HIV/AIDS, cancer, or autoimmune diseases).

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — ID gender
Study Population: Patients diagnosed with generalized chronic periodontitis or gingivitis.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 1970-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Tooth loss rate | From 10 up to 50 years
  Number of teeth lost (initial - final) / number of years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carole CHAKAR, PHD, Study Director — Saint Joseph University of Beirut, Faculty of dental Medicine, Periodontolgy department

IPD SHARING:
Plan to Share IPD: No